CLINICAL TRIAL: NCT03108027
Title: A Randomized, Double-blind, Repeat Dose Cross-over Study to Assess the Bronchodilator Effects of Once Daily QVM149 Following Morning or Evening Dosing for 14 Days Compared to Placebo in Patients With Asthma
Brief Title: Assess Bronchodilator Effect QVM149 Dosed Either in the Morning or Evening Compared to Placebo in Patients With Asthma
Acronym: QVM149
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CQVM149B2209; 2017-000644-17 (EudraCT Number)
Record Dates: First submitted 2017-03-23; First posted 2017-04-11 (Actual); Results first posted 2019-05-21 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2019-05

CONDITIONS: Asthma
Keywords: QVM149,; asthma,; allergic asthma,; allergy triggered asthma,; reactive asthma,; asthma attack,; difficulty breathing
MeSH Terms: conditions — Asthma; Dyspnea

STUDY DESIGN:
Intervention Model Description: This study is to assess the bronchodilator effects of QVM149 dosed once daily either in the morning or in the evening for 2 weeks compared to placebo. It will provide evidence of the comparability of lung function effects of QVM149 irrespective of the administration schedule
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind masking.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence 1 (Experimental): Patients will receive in a sequential order the following interventional treatments: A,B and C.
  Interventions: Drug: Treatment A: Matching placebo (morning dose) and QVM149 150/50/80 μg (evening dose); Drug: Treatment B: QVM149 150/50/80 μg (morning dose) and matching placebo (evening dose); Drug: Treatment C: Placebo (morning dose) and placebo (evening dose)
- Sequence 2 (Experimental): Patients will receive in a sequential order the following interventional treatments: B, A and C.
  Interventions: Drug: Treatment A: Matching placebo (morning dose) and QVM149 150/50/80 μg (evening dose); Drug: Treatment B: QVM149 150/50/80 μg (morning dose) and matching placebo (evening dose); Drug: Treatment C: Placebo (morning dose) and placebo (evening dose)
- Sequence 3 (Experimental): Patients will receive in a sequential order the following interventional treatments: C, B and A.
  Interventions: Drug: Treatment A: Matching placebo (morning dose) and QVM149 150/50/80 μg (evening dose); Drug: Treatment B: QVM149 150/50/80 μg (morning dose) and matching placebo (evening dose); Drug: Treatment C: Placebo (morning dose) and placebo (evening dose)
- Sequence 4 (Experimental): Patients will receive in a sequential order the following interventional treatments : C, A and B.
  Interventions: Drug: Treatment A: Matching placebo (morning dose) and QVM149 150/50/80 μg (evening dose); Drug: Treatment B: QVM149 150/50/80 μg (morning dose) and matching placebo (evening dose); Drug: Treatment C: Placebo (morning dose) and placebo (evening dose)
- Sequence 5 (Experimental): Patients will receive in a sequential order the following interventional treatments: A, C and B.
  Interventions: Drug: Treatment A: Matching placebo (morning dose) and QVM149 150/50/80 μg (evening dose); Drug: Treatment B: QVM149 150/50/80 μg (morning dose) and matching placebo (evening dose); Drug: Treatment C: Placebo (morning dose) and placebo (evening dose)
- Sequence 6 (Experimental): Patients will receive in a sequential order the following interventional treatments: B, C and A.
  Interventions: Drug: Treatment A: Matching placebo (morning dose) and QVM149 150/50/80 μg (evening dose); Drug: Treatment B: QVM149 150/50/80 μg (morning dose) and matching placebo (evening dose); Drug: Treatment C: Placebo (morning dose) and placebo (evening dose)

INTERVENTIONS:
Drug: Treatment A: Matching placebo (morning dose) and QVM149 150/50/80 μg (evening dose) — Matching placebo (morning dose) and QVM149 150/50/80 μg (evening dose)
Drug: Treatment B: QVM149 150/50/80 μg (morning dose) and matching placebo (evening dose) — QVM149 150/50/80 μg (morning dose) and matching placebo (evening dose)
Drug: Treatment C: Placebo (morning dose) and placebo (evening dose) — Placebo (morning dose) and placebo (evening dose)

SUMMARY:
This was a randomized, placebo-controlled, double-blind, six-sequence, three-period cross-over study in asthma patients. The study consisted of a 14-day screening period, followed by a 14-day run-in period, and a treatment epoch which consists of three treatment periods, with a minimum duration of 14 days each followed (for the 2 first treatment periods) by a wash-out period. The duration of each treatment period may be extended up to a duration of 18 days if needed for operational reasons. The third treatment period was followed by a Study Completion evaluation at 1-7 days following the last dose. The treatment periods were separated by wash-out periods of 14 to 21 days duration.

ELIGIBILITY:
Inclusion Criteria:

Patients with a documented physician diagnosis of asthma and who additionally meet the following criteria:

* Patients receiving daily treatment with an inhaled corticosteroid at a low or medium daily dose
* On a stable regimen for at least 4 weeks prior to screening.
* Pre-bronchodilator FEV1 ≥ 60 % and < 100% of the predicted normal value for the patient during screening.
* Patients who demonstrate an increase in FEV1 of ≥ 12 % and ≥ 200 mL after administration of 400 μg salbutamol/360 μg albuterol (or equivalent dose) at Screening. All patients must perform a reversibility test at Screening.
* At screening, and baseline (day 1 pre-dose time) of the first treatment period, vital signs (systolic and diastolic blood pressure and pulse rate) will be assessed in the sitting position and again in the standing position as outlined in the SOM. Sitting and standing vital signs should be within the following ranges:
* oral body temperature between 35.0-37.5 °C
* systolic blood pressure, 90-159 mmHg
* diastolic blood pressure, 50-99 mmHg
* pulse rate, 40-90 bpm
* Hypertensive patients must have been on stable antihypertensive therapy for at least 4 weeks prior to screening to be included in the trial.
* Patients must weigh at least 50 kg at screening to participate in the study, and must have a body mass index (BMI) within the range of 18 to 40 kg/m2.

Exclusion Criteria:

* Contraindicated for treatment with, or having a history of reactions/ hypersensitivity to any of the drugs of a similar class
* Patients who have had an asthma attack/exacerbation requiring systemic steroids or hospitalization or emergency room visit within 1 year of Screening.
* Patients who have had previous intubation for a severe asthma ttack/exacerbation.
* Patients with a history of clinically relevant bronchoconstriction upon repeated forced expiratory maneuvers.
* History of paradoxical bronchospasm in response to inhaled medicines.
* Patients who during the run-in period prior to randomization require the use of ≥12 puffs / 24 hours of rescue medication for 48 hours (over two consecutive days) or who have a decline in PEF from the reference PEFof ≥ 30% for 6 consecutive scheduled PEF readings
* Patients who do not maintain regular day/night, waking/sleeping cycles (e.g., night shift workers).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-06-26 (Actual); Primary Completion 2018-02-24 (Actual); Study Completion 2018-02-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- Germany (5):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Frankfurt Am Main Hessen
  - Novartis Investigative Site, Großhansdorf
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Wiesbaden
- Novartis Investigative Site, Groningen, GZ, Netherlands
- Novartis Investigative Site, Machester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicatrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=413

RESULTS

PARTICIPANT FLOW:
Groups:
- Sequence 1: Patients received in a sequential order the following interventional treatments: A,B and C.
- Sequence 2: Patients received in a sequential order the following interventional treatments: B, A and C.
- Sequence 3: Patients received in a sequential order the following interventional treatments: C, B and A.
- Sequence 4: Patients received in a sequential order the following interventional treatments : C, A and B.
- Sequence 5: Patients received in a sequential order the following interventional treatments: A, C and B.
- Sequence 6: Patients received in a sequential order the following interventional treatments: B, C and A.
Period: Period 1
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 7 | 6 | 6 | 6 | 6 | 6
Completed | 7 | 6 | 6 | 4 | 6 | 6
Not Completed | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Subject/Guardian Decision | 0 | 0 | 0 | 2 | 0 | 0
Period: Period 2
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 7 | 6 | 6 | 4 | 6 | 6
Completed | 7 | 6 | 6 | 4 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Sequence 1 | Sequence 2 | Sequence 3 | Sequence 4 | Sequence 5 | Sequence 6
Started | 7 | 6 | 6 | 4 | 6 | 6
Completed | 7 | 5 | 6 | 4 | 6 | 6
Not Completed | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants randomized to one of six treatment sequences
Arm/Group | All Participants
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.5 (14.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 35
  More than one race | 0
  Unknown or Not Reported | 2

OUTCOME MEASURES:

1. Primary Outcome: FEV1 Standardized Area Under the Curve (AUC 0-24h) After Last Evening Dose of 14-day Treatment Period
Description: Weighted mean forced expiratory volume in 1 second (FEV1) over 24 h (AUC0-24h) following 14 days of treatment with QVM149 dosed in the morning, QVM149 dosed in the evening and placebo.
Time Frame: At the end of each treatment period day 14 pre-dose to 24 hours post-dose.
Population: The pharmacodynamic (PD) analysis set included all patients with any available PD data, who received any dose of study drug and experienced no protocol deviations with relevant impact on PD data.
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- QVM149 am: QVM149 150/50/80 μg o.d. (indacaterol acetate 150 μg/ glycopyrronium bromide 50 μg/ MF 80 μg once daily) administered in the morning (plus matching placebo in the evening)
- QVM149 pm: QVM149 150/50/80 μg o.d. (indacaterol acetate150 μg/ glycopyrronium bromide 50 μg/ MF 80 μg once daily) administered in the evening (plus matching placebo in the morning)
- Placebo: Placebo administered in the morning and in the evening.
Arm/Group | QVM149 am | QVM149 pm | Placebo
Number analyzed (Participants) | 30 | 30 | 33
Liters | 3.4305 (0.15242) | 3.4361 (0.15213) | 2.8209 (0.15259)
Statistical Analysis 1: Comparison: QVM149 am vs Placebo; Test type: Other — A hypothesis test is not planned for this study, inferences are to be performed by interpreting confidence interval of treatment difference.'; Mixed Models Analysis; Mean Difference (Net) = 0.6096, 90% CI 2-sided [0.5380 to 0.6811]
Statistical Analysis 2: Comparison: QVM149 pm vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Mean Difference (Net) = 0.6152, 90% CI 2-sided [0.5437 to 0.6868]
Statistical Analysis 3: Comparison: QVM149 am vs QVM149 pm; Test type: Other — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Mean Difference (Net) = -0.0057, 90% CI 2-sided [-0.0760 to 0.0647]

2. Secondary Outcome: Trough FEV1 After 24h
Description: FEV1 at approximately 24 h after the last p.m. or penultimate a.m. dose. Morning and evening trough FEV1 (L) were analyzed by time of day. For morning trough FEV1 (L) assessments this meant that the spirometric assessment was done approximately 24 h after last morning dose and approximately 12 h after last evening dose.
Time Frame: At the end of each treatment period day 14 pre-dose to 24 hours post-dose.
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QVM149 am | QVM149 pm | Placebo
Number analyzed (Participants) | 35 | 35 | 36
Liters | 3.3731 (0.15037) | 3.4871 (0.15041) | 2.7524 (0.15120)
Statistical Analysis 1: Comparison: QVM149 am vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Mean Difference (Net) = 0.6206, 90% CI 2-sided [0.5335 to 0.7077]
Statistical Analysis 2: Comparison: QVM149 pm vs Placebo; Test type: Other — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Mean Difference (Net) = 0.7347, 90% CI 2-sided [0.6469 to 0.8225]
Statistical Analysis 3: Comparison: QVM149 am vs QVM149 pm; Test type: Other — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Mean Difference (Net) = -0.1141, 90% CI 2-sided [-0.1970 to -0.0311]

3. Secondary Outcome: Peak Expiratory Flow (PEF)
Description: Peak expiratory flow (PEF) is the maximum flow generated during a forceful exhalation, starting from full lung inflationDaily morning and evening peak expiratory flow rate from Day 2 to Day14 during the three treatment periods.
Time Frame: From treatment period start through study completion (up to 19 weeks).
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | QVM149 am | QVM149 pm | Placebo
Number analyzed (Participants) | 35 | 35 | 36
L/min
  Morning average PEF | 489.6 (19.77) | 504.4 (19.78) | 417.5 (19.73)
  Evening average PEF | 522.0 (19.71) | 507.7 (19.71) | 449.0 (19.67)
Statistical Analysis 1: Comparison: QVM149 am vs Placebo; Morning average PEF; Test type: Other — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Mean Difference (Net) = 72.1, 90% CI 2-sided [61.3 to 82.9]
Statistical Analysis 2: Comparison: QVM149 pm vs Placebo; Morning average PEF; Test type: Other — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Mean Difference (Net) = 86.9, 90% CI 2-sided [76.1 to 97.8]
Statistical Analysis 3: Comparison: QVM149 am vs QVM149 pm; Morning average PEF; Test type: Other — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Mean Difference (Net) = -14.8, 90% CI 2-sided [-25.6 to -4.1]
Statistical Analysis 4: Comparison: QVM149 am vs Placebo; Evening average PEF; Test type: Other — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Mean Difference (Net) = 73.1, 90% CI 2-sided [61.9 to 84.2]
Statistical Analysis 5: Comparison: QVM149 pm vs Placebo; Evening average PEF; Test type: Other — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Mean Difference (Net) = 58.7, 90% CI [47.5 to 69.9]
Statistical Analysis 6: Comparison: QVM149 am vs QVM149 pm; Evening average PEF; Test type: Other — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Mean Difference (Net) = 14.4, 90% CI 2-sided [3.3 to 25.5]

ADVERSE EVENTS:
Time Frame: Up to 19 weeks
Groups:
- QVM149 a.m.: QVM149 150/50/80 μg o.d. (indacaterol acetate 150 μg/ glycopyrronium bromide 50 μg/ MF 80 μg once daily) administered in the morning (plus matching placebo in the evening)
- QVM149 p.m.: QVM149 150/50/80 μg o.d. (indacaterol acetate150 μg/ glycopyrronium bromide 50 μg/ MF 80 μg once daily) administered in the evening (plus matching placebo in the morning)
Arm/Group | QVM149 a.m. | QVM149 p.m. | Placebo
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/35 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/35 | 0/36
Other Adverse Events (participants affected / at risk) | 11/35 | 13/35 | 16/36
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QVM149 a.m. (N=35) | QVM149 p.m. (N=35) | Placebo (N=36)
Nasopharyngitis (Infections and infestations) | 2 | 2 | 5
Headache (Nervous system disorders) | 5 | 3 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-03-27): https://cdn.clinicaltrials.gov/large-docs/27/NCT03108027/SAP_000.pdf
  • Study Protocol (2017-03-08): https://cdn.clinicaltrials.gov/large-docs/27/NCT03108027/Prot_001.pdf